CLINICAL TRIAL: NCT01432756
Title: A South African Pilot Worksite Parenting Program to Prevent HIV Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura Bogart, Associate Professor of Pediatrics, Harvard Medical School; Research Director, Division of General Pediatrics, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R34MH090790-02 (NIH); 5R34MH090790 (NIH)
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Parent-Child Relations
Keywords: HIV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list control (No Intervention): Participants in the wait-list control group will not receive the intervention until after the 3-month follow-up assessment.
- Let's Talk Worskite Parenting Program (Experimental): The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
  Interventions: Behavioral: Let's Talk Worksite Parenting Program

INTERVENTIONS:
Behavioral: Let's Talk Worksite Parenting Program — The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
  Arms: Let's Talk Worskite Parenting Program

SUMMARY:
The investigators hypothesize that participants in the worksite parenting program intervention will show significantly better parent-child communication than will participants in the no-treatment (wait-list) control group.

DETAILED DESCRIPTION:
In South Africa, >5 million people, including many adolescents, are living with HIV. Prevalence is increasing throughout South Africa, most precipitously in the Western Cape, the site of our proposed study. The investigators propose to pilot test a multisession worksite-based program to help parents learn how to take an active role in rearing sexually healthy youth. Our specific aims are to: (1) Culturally adapt our US-developed worksite-based program for parents of adolescents to the South African context; (2) Examine whether a worksite-based program for parents of adolescents in South Africa improves the parent-child relationship, including general parent-child communication and communication about sexual health and HIV risk-reduction, as perceived by parents and adolescents; (3) Explore program effects on parents' HIV testing and sexual behaviors; and (4) Explore program effects on theoretically important psychosocial mediators of behavior change (e.g., greater self-efficacy for refusing sex and using condoms, and more perceived disadvantages of unprotected sex). The proposed research is a unique opportunity to adapt and pilot test an innovative HIV prevention intervention that promotes the health of families in a culturally acceptable and sustainable setting.

The research is being conducted in three phases. In Phase 1, the investigators conducted formative qualitative interviews with South African community members who work with adolescents and parents, who work on HIV prevention, and who hold relevant positions at worksites. The investigators used this information from key community members to culturally adapt the program. In Phase 2, the investigators are conducting a process evaluation of one intervention group of 15 parents using qualitative debriefing interviews and quantitative data. In Phase 3, the current phase, the investigators aim to conduct a pilot intervention to refine the program even further and test the evaluation methods with 60 Xhosa and Afrikaans-speaking parents and their 11-15-year-old adolescents (who will participate in the evaluation but not the program). Their outcomes will be compared to a wait-list control group of 60 Xhosa and Afrikaans-speaking parents and their 11-15-year-old adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Parents: Work for City of Cape Town; Are Xhosa-speaking or Afrikaans-speaking; Have a child between the ages of 11-15 (self report); Spend at least 3 days/week with their adolescents
* Children: Eligible if they are between the ages of 11-15 (self report) and have a parent or legal guardian who works in the City of Cape Town who is enrolled in the program.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M. Bogart, PhD, Principal Investigator — Children's Hospital Boston/Harvard Medical School
Locations (1):
- Stellenbosch University, Stellenbosch, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait-list Control - Parent Participants: Parent participants in the wait-list control group will not receive the intervention until after the 3-month follow-up assessment.
- Let's Talk Worskite Parenting Program - Parent Participants: The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
  Let's Talk Worksite Parenting Program: The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence;
- Wait-list Control - Adolescent Partipants: Adolescent wait-list control participants have parents who are in the wait-list control group. Their parents will not receive the intervention until after the 3-month follow-up assessment.
- Let's Talk Worksite Parenting Program - Adolescent Participant: Adolescent participants will have parents who are in the Let's Talk Worksite Parenting Program.
  The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
Period: Overall Study
Arm/Group | Wait-list Control - Parent Participants | Let's Talk Worskite Parenting Program - Parent Participants | Wait-list Control - Adolescent Partipants | Let's Talk Worksite Parenting Program - Adolescent Participant
Started | 32 | 34 | 32 | 34
Completed | 31 | 34 | 30 | 33
Not Completed | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Wait-list Control - Parent Participants: Participants in the wait-list control group will not receive the intervention until after the 3-month follow-up assessment.
- Wait-list Control - Adolescent Participants: Adolescent wait-list control participants have parents who are in the wait-list control group. Their parents will not receive the intervention until after the 3-month follow-up assessment.
- Let's Talk Worksite Parenting Program -Adolescent Participants: Adolescent participants will have parents who are in the Let's Talk Worksite Parenting Program.
  The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
- Total: Total of all reporting groups
Arm/Group | Wait-list Control - Parent Participants | Let's Talk Worskite Parenting Program - Parent Participants | Wait-list Control - Adolescent Participants | Let's Talk Worksite Parenting Program -Adolescent Participants | Total
Number analyzed (Participants) | 32 | 34 | 32 | 34 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 32 | 34 | 66
  Between 18 and 65 years | 32 | 34 | 0 | 0 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 16 | 13 | 53
  Male | 20 | 22 | 16 | 21 | 79
Region of Enrollment [Number; unit: participants]
  South Africa | 32 | 34 | 32 | 34 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Topics Discussed Between Parent and Child
Description: Measured using the Parent-Child Communication Scale (communication on sexual and HIV topics that the intervention covers) for both parent and child participants in pre- and post-assessments. This is a measurement of the number of sex and HIV topics discussed. 16 topics were assessed, including how women get pregnant, how to use condoms to prevent pregnancy and HIV, and how to recognize sexual pressure.
  For each topic, participants answered yes or no if they discussed it, and then rate between 1-16 to indicate their communication (higher scores mean better communication). The total scores is reported as the sum of the 16 items, and can range from 0-16.
Time Frame: 6 months
Population: Each dyad consisted of one parent and their adolescent child. Sixty-six parents and 66 adolescents participated.
Measure: Mean (Standard Deviation); unit: number of sex and HIV topics discussed
Arm/Group | Wait-list Control - Parent Participants | Let's Talk Worskite Parenting Program - Parent Participants | Wait-list Control - Adolescent Participants | Let's Talk Worksite Parenting Program -Adolescent Participants
Number analyzed (Participants) | 32 | 34 | 32 | 34
number of sex and HIV topics discussed
  Baseline | 8.3 (5.7) | 7.8 (4.8) | 9.4 (4.0) | 7.2 (4.7)
  First Follow-up | 9.3 (5.7) | 12.4 (4.3) | 9.2 (5.1) | 9.2 (4.8)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Let's Talk Worskite Parenting Program: The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence; and alcohol/substance use. Parent participants will receive weekly exercises to help them practice their new skills at home with their child.
  Let's Talk Worksite Parenting Program: The Let's Talk Worksite Parenting Program is designed for Xhosa-speaking and Afrikaans speaking parents (separate sessions) with 11- to 15-year-old children. The 5-session program meets weekly for 2 hours. The program will include instruction on parenting skills and will cover topics relevant to promoting adolescent sexual health, such as; parental involvement; adolescent sexual behavior; HIV; violence;
Arm/Group | Wait-list Control | Let's Talk Worskite Parenting Program
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/68
Other Adverse Events (participants affected / at risk) | 0/64 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes